CLINICAL TRIAL: NCT02667808
Title: Exploring the Impact of HIV and ART on Knowledge, Attitudes and Practices in Reproductive Health in Lilongwe, Malawi
Acronym: HIV KAP
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Lisa Haddad, Assistant Professor, Emory University
Other Study IDs: IRB00051780
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-01

CONDITIONS: HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Focus Group: Participants with HIV and receiving antiretroviral therapy (ART) will participate in four to eight group discussions aimed to evaluate fertility intentions, family planning, and sexual health behaviors. Discussions will be 1-2 hours in length. Groups will be conducted among men and women.
  Interventions: Other: Focus Group
- Questionnaire: Participants with HIV will complete a questionnaire assessing reproductive health knowledge, attitudes and practices related to family planning, and fertility and sexual health. The questionnaire will take no longer than 30 minutes to complete.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Focus Group — Subjects will participate in four to eight group discussions aimed to evaluate fertility intentions, family planning, and sexual health behaviors. Discussions will be 1-2 hours in length. Groups will be conducted among men and women.
  Groups: Focus Group
Other: Questionnaire — Participants will complete a questionnaire assessing reproductive health knowledge, attitudes and practices related to family planning, and fertility and sexual health. The questionnaire will take no longer than 30 minutes to complete.
  Groups: Questionnaire

SUMMARY:
The aim of this study is to identify reproductive health priorities among individuals living with HIV.This study also seeks to explore factors that influence fertility, family planning, and sexual behavior among individuals with HIV who are receiving antiretroviral therapy (ART).

DETAILED DESCRIPTION:
The aim of this study is to identify reproductive health priorities among individuals living with HIV.This study also seeks to explore factors that influence fertility, family planning, and sexual behavior among individuals with HIV who are receiving antiretroviral therapy (ART).

This is a mixed method study in which subjects will participate in focused group discussions and complete a questionnaire. Discussions will be 1-2 hours in length aimed to evaluate fertility intentions, family planning, and sexual health behaviors. Data collected from the focus groups will be analyzed for common themes to generate questionnaires to assess reproductive health knowledge, attitudes and practices related to family planning, and fertility and sexual health among persons living with HIV.

ELIGIBILITY:
Focus Group Arm

Inclusion Criteria:

* Client registered at either of the participating Lighthouse clinics (Kamuzu Central Hospital (KCH) or Bwaila Hospital)
* On antiretroviral treatment (ART) for the past 6 months
* Sexually active within the past 6 months
* HIV positive

Exclusion Criteria:

No exclusion criteria specified

Questionnaire Arm

Inclusion Criteria:

* Client registered at either of the participating Lighthouse clinics (Kamuzu Central Hospital (KCH) or Bwaila Hospital)
* Sexually active within the past 6 month
* HIV positive

Exclusion Criteria:

No exclusion criteria specified

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Persons living with HIV in Lilongwe, Malawi recruited from The Lighthouse Trust Clinic
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Perception of ideal family size assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Perception of ideal family size will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Perception of social pressures regarding fertility intentions assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Perception of social pressures regarding fertility intentions will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Perception of familial pressures regarding fertility intentions assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Perception of familial pressures regarding fertility intentions will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Perception of partner pressures regarding fertility intentions assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Perception of partner pressures regarding fertility intentions will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Influence of human immunodeficiency virus (HIV) on fertility intentions assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Influence of human immunodeficiency virus (HIV) on fertility intentions will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Influence of antiretroviral therapy (ART) on fertility intentions assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Influence of antiretroviral therapy (ART) on fertility intentions will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Perception of concordance among couples on fertility intention assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  The agreement on fertility intention among couples will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Perception of how relationship status influences fertility intentions assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  The perception of how relationship status influences fertility intentions will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Perception of how reproductive health issues impact fertility intentions assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Perception of how reproductive health issues impact fertility intentions will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Knowledge regarding family planning methods assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Knowledge regarding family planning methods will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Knowledge regarding family planning misconceptions assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Knowledge regarding family planning misconceptions and beliefs will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Current family planning methods assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Current family planning methods will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Previously used family planning methods assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Previously used family planning methods will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Intent to use family planning methods assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Intent to use family planning methods will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Perception of social influence on family planning methods assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Perception of social influence on family planning methods will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Perception of familial influence on family planning methods assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Perception of familial influence on family planning methods will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Perception of partner influence on family planning methods assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Perception of partner influence on family planning methods will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Human immunodeficiency virus (HIV) influence on family planning methods assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Human immunodeficiency virus (HIV) influence on family planning methods will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Antiretroviral therapy (ART) use influence on family planning methods assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Antiretroviral therapy (ART) use influence on family planning methods will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours
Antiretroviral therapy (ART) non-use influence on family planning methods assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Antiretroviral therapy (ART) non-use influence on family planning methods will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Influence of human immunodeficiency virus (HIV) on use of dual protection assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Influence of HIV on use of dual protection will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Influence of human immunodeficiency virus (HIV) on non-use of dual protection assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Influence of HIV on non-use of dual protection will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Influence of antiretroviral therapy (ART) on use of dual protection assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Influence of ART on use of dual protection will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Influence of antiretroviral therapy (ART) on non-use of dual protection assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Influence of ART on non-use of dual protection will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Perception of sexually transmitted infection (STI) risk assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Perception of sexually transmitted infection (STI) risk will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.
Perception of risk of human immunodeficiency virus (HIV) transmission to partners or children assessed by focus group discussion | Discussion Visit (Day 0, Up to 2 hours)
  Perception of risk of HIV transmission to partners or children will be discussed in a focus group setting between 6-8 men or women. Focus groups will be facilitated by a trained member of the research team. The discussions will be audio taped and there will be a note-taker attending each group. Notes will be taken during the groups should elements of the audio recording need clarification as well as to capture non-verbal responses and communication. Focus group discussion will take between one to two hours.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Haddad, MD, Principal Investigator — Emory University
Locations (1):
- The Lighthouse Trust, Lilongwe, Malawi